CLINICAL TRIAL: NCT06839937
Title: A Virtual Reality Couples' Intervention for Sexual Victimization Prevention: a Gender-swapping Transformative Approach (REVISE)
Brief Title: A Virtual Reality Couples' Intervention for Sexual Victimization Prevention: a Gender-swapping Transformative Approach
Acronym: REVISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Oberta de Catalunya (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government); European Social Fund (Other)
Responsible Party: Principal Investigator, Adrián Montesano, Associate Professor and Principal Investigator, Universitat Oberta de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCIN/AEI/10.13039/501100011033; PID2022-141198OB-I00 (Other Grant/Funding Number: MCIN/AEI/10.13039/501100011033 & FSE+)
Record Dates: First submitted 2025-02-05; First posted 2025-02-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Sexual Harassment; Gender Based Violence; Empathy; Virtual Reality Exposure Therapy
Keywords: Sexual Harassment; Gender-Based Violence; Immersive Virtual Reality; Violence Prevention; Sexism; VR Intervention; Violence Against Woman
MeSH Terms: conditions — Sexual Harassment; Sexism

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three independent intervention groups:
  1. Identity Exchange with Exposure to Sexual Harassment: Male participants will embody their female partner's avatar in a VR harassment scenario.
  2. Identity Exchange without Harassment Exposure: Male participants will embody their female partner's avatar in a neutral VR scenario.
  3. Third-person Observer Condition: Male participants will observe a harassment scenario in VR without identity exchange.
  Each participant remains in their assigned condition throughout the study, and comparisons are made between groups based on empathy, gender attitudes, and harassment-related responses.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Identity Exchange with Exposure to Sexual Harassment (Experimental): Participants will experience a virtual reality (VR) perspective-taking intervention in which they embody their female partner's avatar in a scenario depicting sexual harassment. This immersive experience aims to enhance empathy and reduce the acceptance of sexual harassment. Physiological responses (eye tracking and pupillometry) will be recorded, and participants will complete pre- and post-intervention self-reports.
  Interventions: Behavioral: REVISE - Virtual Reality Gender-Swap with Harassment Exposure
- Identity Exchange without Harassment Exposure (Experimental): Participants will embody their female partner's avatar in a neutral VR scenario without any harassment. This condition serves to evaluate the effects of identity exchange alone, without exposure to gender-based violence, on empathy and gender attitudes. Pre- and post-intervention assessments and physiological measures will be collected.
  Interventions: Behavioral: REVISE - Virtual Reality Gender-Swap without Harassment
- Third-Person Observer Condition (No Intervention): Participants will observe a VR scenario depicting sexual harassment from a third-person perspective, without experiencing identity exchange. This condition acts as a control to determine whether passive observation differs from immersive perspective-taking in modifying attitudes toward gender-based violence. Self-reports and physiological responses will be also analyzed.

INTERVENTIONS:
Behavioral: REVISE - Virtual Reality Gender-Swap with Harassment Exposure — Participants will embody a virtual avatar of their female partner in a sexual harassment scenario using full-body tracking, and identity exchange in virtual reality (VR). The goal is to assess whether experiencing harassment from a first-person perspective increases empathy and decreases tolerance toward sexual harassment.
  Arms: Identity Exchange with Exposure to Sexual Harassment
Behavioral: REVISE - Virtual Reality Gender-Swap without Harassment — Participants will embody a virtual avatar of their female partner in a neutral social interaction scenario using VR-based identity exchange. This condition controls for the effect of perspective-taking alone, without exposure to harassment, to evaluate its impact on empathy and gender attitudes.
  Arms: Identity Exchange without Harassment Exposure

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of REVISE (REalidad Virtual Inmersiva y SExualidad), an immersive virtual reality (IVR) intervention designed to promote empathy and reduce sexual harassment behaviors in heterosexual cisgender men.

The main questions that this study aims to answer are as follows.

Does experiencing gender swapping in IVR increase empathy towards survivors of sexual harassment?

Does the intervention modify attitudes toward gender roles and sexual harassment?

Researchers will compare the three experimental groups to evaluate the effects of IVR:

1. Identity Exchange Group with Exposure to Sexual Harassment: Participants embodied their partner's identity in a VR harassment scenario.
2. Identity Exchange Group without Harassment Exposure: Participants embodied their partner's identity in a neutral VR scenario.
3. Third-person Observer Group: Participants observe a harassment scenario in VR from their own perspective.

Participants will:

1. Attend one virtual reality session in a laboratory setting.
2. Undergo pre- and post-intervention assessments and a three-month follow-up.
3. Complete self-report questionnaires and physiological measures (eye tracking and pupillometry).
4. Participate in semi-structured interviews about their experiences. This study aims to explore how immersive VR embodiment can be used as a tool for gender violence prevention by fostering perspective-taking and behavioral change.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) designed to evaluate the efficacy of REVISE (REalidad Virtual Inmersiva y SExualidad), an immersive virtual reality (IVR) intervention, to promote empathy and reduce sexual harassment behaviors in heterosexual cisgender men. This study will assess whether experiencing sexual harassment from a first-person perspective using IVR embodiment techniques can lead to changes in attitudes and behaviors related to gender roles and sexual violence.

Study Design

* Design: Randomized controlled trial (RCT) with a 1:1:1 allocation ratio.
* Population: 90 heterosexual cisgender couples (180 participants) aged 18-39 years.
* Study Setting: This study will be conducted in a controlled laboratory environment at the Interdisciplinary Research and Innovation Hub of the Universitat Oberta de Catalunya (UOC), equipped with advanced VR and physiological tracking technologies.
* Conditions:

  1. Identity Exchange with Exposure to Sexual Harassment (Experimental Condition 1)
  2. Identity Exchange without Harassment Exposure (Experimental Condition 2) 3. Third-person Observer Condition (Control Group)
* Intervention Duration: One VR session (~60 minutes) with pre- and post-intervention assessments and a three-month follow-up.

Intervention Procedures

1. Pre-intervention assessment

   * Participants complete self-report questionnaires measuring empathy, gender role attitudes, and harassment perceptions.
   * Baseline physiological measures (eye tracking and pupillometry) are recorded. - Participants are assigned to one of the three conditions.
2. VR Intervention:

   * Participants undergo a mirror embodiment task to establish a sense of virtual body ownership.
   * The male participant embodies his female partner's avatar in a VR scenario (conditions 1 and 2).
   * Participants experience the designated VR scenario (harassment, neutral, or observational).
   * Physiological responses are collected in real time.
3. Post-intervention assessment

   * Participants complete self-report measures to assess changes in empathy and gender attitudes.
   * Physiological data analysis (pupil dilation and eye gaze fixation) is conducted. - Semi-structured interviews explore subjective experiences.
4. Three-month follow-up:

   * Participants complete longitudinal measures to assess sustained behavioral and attitudinal changes.

Outcome Measures

1. Primary Outcome: Change in empathy scores (Interpersonal Reactivity Index). 2. Secondary Outcomes:

* Gender role attitudes (Ambivalent Sexism Inventory).
* Dyadic relationship quality and flourishing
* Harassment-related attitudes - Eye-tracking and pupillometry responses during VR.
* Qualitative insights from the post-intervention interviews.

Sample Size Justification A sample of 90 couples (180 individuals) was determined based on an estimated effect size of d = 0.5, an alpha risk of 0.05, and a power of 0.86. Participants will be randomized using block randomization (block sizes of 3 or 6) to ensure balance across the conditions.

Data Management and Quality Assurance

1. Data Collection

   * Self-reported data will be collected using secure online survey tools.
   * Physiological data will be automatically recorded using VR-compatible eye-tracking and pupillometry systems.
2. Data Validation and Security

   * The dataset will undergo automatic range checks to detect anomalies.
   * Double data entry procedures will be implemented for self-report responses.
   * Only authorized researchers will have access to identifiable data, stored on encrypted servers.
3. Missing Data Handling:

   * Missing values will be addressed using multiple imputation techniques.
   * Sensitivity analyses will be conducted to determine the impact of the missing data.

Statistical Analysis Plan

1. Primary Analysis:

   - Repeated measures ANOVA will assess within- and between-group differences in empathy scores over time.
2. Secondary Analyses:

   * Generalized Estimating Equations (GEE) will model longitudinal changes in gender attitudes.
   * Mixed-effects models will analyze physiological responses (eye tracking and pupil dilation).
   * Qualitative data from the interviews will be subjected to thematic analysis using NVivo software.

Ethical Considerations

* The study has received approval from the Research Ethics Committee of the Universitat Oberta de Catalunya.
* Participants will provide informed consent prior to participation.
* Psychological debriefing and support resources will be available to participants.

Dissemination Plan

The findings will be as follows:

* Peer-reviewed journal publications.
* Academic conferences in psychology, gender studies, and VR research.
* Open science repositories for data transparency.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 39 years old.
* Couples must have been in a romantic relationship for at least six months.
* Both partners must provide explicit informed consent to participate.
* Participants must be able to read and write in Spanish to ensure comprehension of the study materials.

Exclusion Criteria:

* Individuals with any physical condition that may hinder the use of VR equipment (e.g., epilepsy or severe motion sickness).
* Individuals with a history of sexual harassment or problematic substance use, including drug or alcohol abuse.
* Individuals experiencing significant mental health difficulties that require intensive treatment.
* Participants with prior exposure to similar VR-based gender perspective-taking interventions.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is open to heterosexual cisgender couples, where the male partner identifies as cisgender man and the female partner identifies as cisgender woman. Both partners must be in a romantic relationship at the time of participation. Individuals who identify as non-binary, transgender, or gender non-conforming are not eligible for this study, as the intervention specifically focuses on gender-based perspective-taking between cisgender men and women.
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Empathy Scores (Interpersonal Reactivity Index - IRI) | Baseline, immediately post-intervention, 3-month follow-up
  Empathy will be assessed using the Interpersonal Reactivity Index (IRI), a validated self-report measure that evaluates different components of empathy, including perspective-taking and empathic concern. The IRI consists of 28 items, each rated on a 5-point Likert scale (0 = Does not describe me well to 4 = Describes me very well). The total score ranged from 0 to 112, with higher scores indicating greater levels of empathy. Cronbach's alpha ranged from .68 to .80. Participants will complete the IRI at baseline (pre-intervention), immediately post-intervention, and at a three-month follow-up to assess changes over time. Higher scores indicate greater empathy levels.

SECONDARY OUTCOMES:
Change in Gender Role Attitudes (Ambivalent Sexism Inventory - ASI) | Baseline, immediately post-intervention, 3-month follow-up
  Gender role attitudes will be measured using the Ambivalent Sexism Inventory (ASI), which assesses two factors: hostile and benevolent sexism. We will use the brief version composed of 12 items (6 items in each factor) with Cronbach's alphas of .75 and .81. Higher scores indicate greater sexist attitudes. Participants will complete the ASI at baseline, post-intervention, and 3-month follow-up to evaluate changes in gender-related beliefs.
Change in Communication Patterns (Communication Patterns Questionnaire - CPQ) | Baseline, immediately post-intervention, 3-month follow-up
  Communication patterns in close relationships will be assessed using the Spanish version of the Communication Patterns Questionnaire (CPQ). The CPQ is a self-report measure that evaluates three dimensions of communication: mutual constructive communication, communication avoidance or demand/withdrawal, and aggressive communication. Participants will complete the CPQ at baseline (pre-intervention), immediately post-intervention, and at a three-month follow-up to assess changes in communication styles over time. The questionnaire consists of 24 items, each rated on a 9-point Likert scale ranging from 1 ("Very unlikely") to 9 ("Very likely"). Higher scores indicate greater use of the corresponding communication strategy. Cronbach alpha in Spain ranged from .62 to .84.
Change in Relationship Satisfaction (Dyadic Adjustment Scale - DAS) | Baseline, immediately post-intervention, 3-month follow-up
  We will use the Spanish brief version of the DAS. It is composed of 13 items answered in a variable Likert scale and those items are grouped under three second order factors and one of first order structure. The scale in its short form presents a cut-off of 44. The higher the score the best adjustment is observed. Cronbach alpha was .83.
Change in Couple Flourishing (Couple Flourishing Measure - CFM) | Baseline, immediately post-intervention, 3-month follow-up
  Couple flourishing will be assessed using the Couple Flourishing Measure (CFM), a unidimensional self-report instrument. The Spanish validated version by Saavedra-Roa et al. will be used in this study. Participants will complete the CFM at baseline (pre-intervention), immediately post-intervention, and at a three-month follow-up to assess changes in relationship satisfaction and flourishing over time. The questionnaire consists of 16 items, each rated on a 7-point visual analogue Likert scale ranging from 1 (Distressed relationship), 4 (Satisfied relationship), to 7 (Flourishing relationship). The total score ranges from 16 to 112, with higher scores indicating greater couple flourishing. The instrument demonstrated high internal consistency reliability (α = .94).
Change in Acceptance of Modern Myths about Sexual Aggression (AMMSA Scale) | Baseline, immediately post-intervention, 3-month follow-up
  Attitudes towards modern myths about sexual aggression will be assessed using the Acceptance of Modern Myths about Sexual Aggression Scale (AMMSA; Gerger et al., 2007). The Spanish adapted and validated version (Megías et al., 2011) will be used in this study. The AMMSA is a self-report measure designed to evaluate subtle beliefs that justify or minimize sexual aggression. Participants will complete the AMMSA at baseline (pre-intervention), immediately post-intervention, and at a three-month follow-up to assess changes in the acceptance of sexual aggression myths over time. The questionnaire consists of 30 items, each rated on a 7-point Likert scale, ranging from 1 ("Totally disagree") to 7 ("Totally agree"). Higher scores indicate greater acceptance of modern myths about sexual aggression. Cronbach alpha in a Spanish sample was .91.
Change in Body Ownership Illusion | During VR exposure at two assessment points: (1) Mirror embodiment phase (approximately 5 minutes after VR start) and (2) Farewell phase (at the end of VR exposure, approximately 15 minutes after VR start).
  Body ownership illusion will be assessed to measure the extent to which participants experience the illusion of embodying their self-avatar and their partner's avatar. This measure evaluates embodiment and agency from a first-person perspective during the VR experience. A validated four-item scale will be administered verbally in two phases: (1) mirror embodiment with the assistant and (2) farewell with the assistant . In the first phase, the assistant will instruct the participant to look into a virtual mirror and ask: "On a scale from 0 to 10, to what extent did you feel that the virtual body in the mirror was your own?" and "When looking down, did you feel that the virtual body was yours?" In the second phase, the assistant will ask: "Did you feel that you owned a different body?" and "Did you feel fear of aggression?" Higher scores indicate a stronger experience of embodiment.
Change in Physiological Arousal (Pupillometry) | From the start of VR exposure until the completion of the VR session (approximately 15 minutes). Data will be collected in real-time during this period.
  Physiological arousal will be measured using pupillometry, which records minute fluctuations in the pupil diameter in response to stimuli. Pupil dilation is an indicator of autonomic nervous system activation, and greater pupil dilation is associated with negative emotional processing. The key metric recorded will be pupil diameter ratio (measured in millimeters): the relative change in pupil size in response to VR stimuli. The pupil data will be sampled at a minimum frequency of 60 Hz with a visual angle accuracy of 0.5°. Artifacts such as pupil amplitude outliers (<1 mm or >9 mm), drifts, and blinks will be coded as missing values. A 10 Hz low-pass filter will be applied to smooth the data.
Change in Visual Attention (Eye-Tracking Data) | From the start of VR exposure until the completion of the VR session (approximately 15 minutes). Data will be collected in real-time during this period.
  Visual attention will be assessed using eye tracking technology integrated into VR goggles. Eye tracking measures fixation behavior as an indicator of attention allocation toward erotic stimuli, based on sexual objectification theory (Hollett et al., 2022). Two key parameters will be recorded: 1) fixation count (measured in number of fixations): number of available fixations on a specified area of interest (VR model's neckline) and dwell time (measured in milliseconds), and total duration of fixations on the area of interest (neckline). Fixation was defined as a continuous gaze lasting at least 100 ms.
Changes in affective responses | During VR exposure at one assessment point: Farewell phase (at the end of VR exposure, approximately 15 minutes after VR start).
  Self-Assessment Manikin (SAM) will be used to assess participants' affective responses during the intervention. This is a non-verbal, pictorial scale that evaluates three dimensions of emotional reaction: Valence (from negative/unpleasant to positive/pleasant), Arousal (from calm to excited), and Dominance (from feeling dominated to feeling in control). Each dimension is rated on a 9-point scale: 1 indicates the lowest intensity (e.g., unpleasant, calm, or dominated), and 9 indicates the highest intensity (e.g., pleasant, excited, or dominant). Higher scores represent more positive emotional valence, higher arousal, and greater sense of control or dominance
Qualitative Insights from Participant Experience | Immediately post-intervention
  Participants will complete semi-structured interviews post-intervention to explore their experiences and perceptions of the VR embodiment task. Interviews will be transcribed and analyzed using thematic analysis to identify key themes related to empathy, gender role reflection, and perceived impact of the intervention.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of privacy and confidentiality concerns, as the study involves sensitive topics related to sexual harassment and gender identity. Given the nature of the intervention and the potential risk of re-identification, all collected data will be stored securely and will only be accessible to the research team in accordance with institutional ethical guidelines and data protection regulations (e.g., GDPR). Aggregated results will be published in peer-reviewed journals, but the raw participant-level data will remain confidential.

REFERENCES:
- [Background] Carvalho J, Rosa PJ, Pereira B. Dynamic Risk Factors Characterizing Aggressive Sexual Initiation by Female College Students. J Interpers Violence. 2021 Mar;36(5-6):2455-2477. doi: 10.1177/0886260518760010. Epub 2018 Mar 5. PMID 29502500
- [Background] Hollett RC, Rogers SL, Florido P, Mosdell B. Body Gaze as a Marker of Sexual Objectification: A New Scale for Pervasive Gaze and Gaze Provocation Behaviors in Heterosexual Women and Men. Arch Sex Behav. 2022 Aug;51(6):2759-2780. doi: 10.1007/s10508-022-02290-y. Epub 2022 Mar 29. PMID 35348918
- [Background] Bradley MM, Lang PJ. Measuring emotion: the Self-Assessment Manikin and the Semantic Differential. J Behav Ther Exp Psychiatry. 1994 Mar;25(1):49-59. doi: 10.1016/0005-7916(94)90063-9. PMID 7962581
- [Background] Ventura S, Cardenas G, Miragall M, Riva G, Banos R. How Does It Feel to Be a Woman Victim of Sexual Harassment? The Effect of 360 degrees -Video-Based Virtual Reality on Empathy and Related Variables. Cyberpsychol Behav Soc Netw. 2021 Apr;24(4):258-266. doi: 10.1089/cyber.2020.0209. Epub 2020 Oct 20. PMID 33085513
- [Background] Jouriles EN, McDonald R, Kullowatz A, Rosenfield D, Gomez GS, Cuevas A. Can virtual reality increase the realism of role plays used to teach college women sexual coercion and rape-resistance skills? Behav Ther. 2009 Dec;40(4):337-45. doi: 10.1016/j.beth.2008.09.002. Epub 2008 Oct 31. PMID 19892079
- [Background] Riva G, Banos RM, Botella C, Mantovani F, Gaggioli A. Transforming Experience: The Potential of Augmented Reality and Virtual Reality for Enhancing Personal and Clinical Change. Front Psychiatry. 2016 Sep 30;7:164. doi: 10.3389/fpsyt.2016.00164. eCollection 2016. PMID 27746747
- [Background] Maister L, Slater M, Sanchez-Vives MV, Tsakiris M. Changing bodies changes minds: owning another body affects social cognition. Trends Cogn Sci. 2015 Jan;19(1):6-12. doi: 10.1016/j.tics.2014.11.001. Epub 2014 Dec 15. PMID 25524273
- [Background] Dobbin F, Kalev A. The promise and peril of sexual harassment programs. Proc Natl Acad Sci U S A. 2019 Jun 18;116(25):12255-12260. doi: 10.1073/pnas.1818477116. Epub 2019 Jun 3. PMID 31160444
- [Background] DeGue S, Valle LA, Holt MK, Massetti GM, Matjasko JL, Tharp AT. A systematic review of primary prevention strategies for sexual violence perpetration. Aggress Violent Behav. 2014 Jul-Aug;19(4):346-362. doi: 10.1016/j.avb.2014.05.004. PMID 29606897
- [Background] Gunarathne L, Bhowmik J, Apputhurai P, Nedeljkovic M. Factors and consequences associated with intimate partner violence against women in low- and middle-income countries: A systematic review. PLoS One. 2023 Nov 8;18(11):e0293295. doi: 10.1371/journal.pone.0293295. eCollection 2023. PMID 37939106
- [Background] Tourne Garcia M, Herrero Velazquez S, Garriga Puerto A. [Health consequences of violence against women by the couple]. Aten Primaria. 2024 Nov;56(11):102903. doi: 10.1016/j.aprim.2024.102903. Epub 2024 Mar 27. Spanish. PMID 38538482